CLINICAL TRIAL: NCT06378970
Title: Effects of Audio Book Application on Anxiety and Vital Signs With Patients Who Receive NIMV Support
Brief Title: Audio Books Effects on Anxiety and Vital Sings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Esra Oksel, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1T/49
Record Dates: First submitted 2024-04-06; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Non-invasive Mechanical Ventilation
Keywords: respiration support; anxiety; vital signs; audio book
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio Book Application Group (Experimental): Patients were made to listen to audio books.
  Interventions: Other: Audio Book Application
- Control Group (No Intervention): No Intervention

INTERVENTIONS:
Other: Audio Book Application — The Audio Book Application Preference Form asked about book preferences other than horror and thriller genres. The selected audiobook was played with headphones via tablet/smartphone. Separate headphones were used for each patient. Patient Follow-up Form and Facial Anxiety Scale evaluations; the initial measurement (M0) was evaluated before the intervention, the first measurement (M1) at the 15th minute of the intervention, the second measurement (M2) at the 30th minute of the intervention, and the third measurement (M3) 30 minutes after the end of the intervention. Care was taken to ensure that there was no deterioration in the comfort of individuals due to the intervention. In the selection of audio books, language fluency, spelling rules and accessibility were taken into consideration and audiobook platforms to which the researchers were members were used.
  Arms: Audio Book Application Group

SUMMARY:
Objectives: This study aimed to investigate the effect of audio book use on anxiety and vital signs in patients receiving non-invasive mechanical ventilation (NIMV) support.

Research Methodology/Design: It is an experimental-randomised controlled study. Settings: The study was carried out with patients hospitalised in the Chest Diseases Intensive Care Unit of a university hospital and NIMV support. The participants consisted of 60 people, 30 in the intervention group and 30 in the control group. Before starting the application in the intervention group, the book preferences of the patients were determined and the selected audio book was played to the patients with headphones via tablet/smartphone. No additional application was made to the control group.

Main Outcome Measures: Anxiety levels and vital signs in the intervention group were evaluated before, 15 minutes, 30 minutes and 30 minutes after the end of the intervention. In the control group, only routine care continued and anxiety levels, and vital signs were assessed simultaneously with the intervention group.

DETAILED DESCRIPTION:
Noninvasive mechanical ventilation (NIMV) is a method that provides positive-pressure respiratory support through a mask without the use of an endotracheal tube. In patients in intensive care units, various symptoms such as agitation, anxiety, and disorientation occur due to factors like constant monitoring, limited movement, painful interventions, intensive treatment protocols, and lack of information. Increased anxiety can result in the rejection of NIMV and may lead to unfavorable outcomes, including treatment failure and prolonged hospitalization.

Objectives: It is crucial to manage anxiety and monitor the resulting changes in vital signs in patients receiving NIMV support. In this context, distraction techniques can be employed by nurses to alleviate anxiety and enhance patient compliance with NIMV therapy. This study aimed to investigate the potential of audio books as a distraction technique to reduce anxiety and stabilize vital signs in patients undergoing NIMV support.

Study Design and Setting: The study employed an experimental-randomized controlled design. It was conducted with patients hospitalized in the Chest Diseases Intensive Care Unit of a university hospital who were receiving NIMV support.

Participants: The study sample consisted of 60 patients, with 30 assigned to the intervention group and 30 to the control group. To account for potential losses during the research process, the number of participants was increased by 25% above the minimum required sample size, setting the minimum sample size per group at 30 patients. Participants were numbered sequentially based on their hospital admission.

Intervention: Before initiating the intervention, the audio book preferences of the patients in the intervention group were determined. The selected audio book was played to the patients using headphones through a tablet or smartphone. No additional interventions were applied to the control group, which received only routine care.

Outcome Measures: Anxiety levels and vital signs were assessed at four different time points in the intervention group: before the intervention, 15 minutes, 30 minutes, and 30 minutes after the end of the intervention. In the control group, anxiety levels and vital signs were assessed concurrently with the intervention group.

Data Analysis: The collected data were analyzed using descriptive statistics, including number and percentage distributions. For comparative analyses between groups, the Mann Whitney U Test, Chi-Square Test, Independent Sample t Test, Friedman Test, One-Way Analysis of Variance, Wilcoxon Test, and Bonferroni Posthoc Test were employed.

ELIGIBILITY:
Inclusion Criteria:

* Not having been diagnosed with a neurological disease.
* At least 6 hours have passed since admission to intensive care
* Being administered NIMV at least once after admission to intensive care
* Not having taken any action that would increase anxiety at least 2 hours before the use of NIMV
* Using an ora-nasal mask
* Not having been diagnosed with a psychiatric disease
* Not having sedation treatment
* Being hemodynamically stable
* No hearing problems
* Agreeing to participate in the research

Exclusion Criteria:

* Refusing to participate in the research
* Using a full face mask
* Having deteriorated general condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Facial Anxiety Scale | before intervention, 15th minute of intervention, 30th minute of intervention 30 minute after intervention
  The Facial Anxiety Scale is a measurement tool in which patients self-report their anxiety levels. It consists of five face shapes, the leftmost face expression indicates the absence of anxiety, while the level of anxiety increases towards the right (scored between 1-5). According to the Faces Anxiety Scale, a score of 3 and above by patients indicates that the level of anxiety is at medium and high levels the Faces Anxiety Scale is a valid means of measuring anxiety in intensive care patients.
Patient Follow-up Form | before intervention, 15th minute of intervention, 30th minute of intervention 30 minute after intervention
  It was prepared by the researcher. Haemodynamic parameters including systolic diastolic blood pressure, pulse rate, respiratory rate and oxygen saturation were included.
Audio Book Application Preference Form | 4 month
  It was prepared by the researchers.there are questions about the preferred book, listening time.
Patient Information Form | 4 month
  There are a total of 7 questions in the patient introduction form, including 4 questions on the socio-demographic characteristics of the patients (age, sex, education level, marital status) and 3 questions on the diagnosis of health status (diagnosis of hospitalisation, presence of chronic disease in addition to the diagnosis of hospitalisation, number of days of NIMV connection).

CONTACTS AND LOCATIONS:
Overall Officials: Esra OKSEL, PhD, Study Director — Ege University
Locations (1):
- Ege University, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKinley S, Coote K, Stein-Parbury J. Development and testing of a Faces Scale for the assessment of anxiety in critically ill patients. J Adv Nurs. 2003 Jan;41(1):73-9. doi: 10.1046/j.1365-2648.2003.02508.x. PMID 12519290
- [Background] McKinley S, Stein-Parbury J, Chehelnabi A, Lovas J. Assessment of anxiety in intensive care patients by using the Faces Anxiety Scale. Am J Crit Care. 2004 Mar;13(2):146-52. PMID 15043242
- [Background] Iyigun E, Pazar B, Tastan S. A study on reliability and validity of the Turkish version of the Face Anxiety Scale on mechanically-ventilated patients. Intensive Crit Care Nurs. 2016 Dec;37:46-51. doi: 10.1016/j.iccn.2016.05.002. Epub 2016 Jul 9. PMID 27401047